CLINICAL TRIAL: NCT06728644
Title: The Safety and Efficacy of L-arginine in Patients With Polycystic Ovary Syndrome
Brief Title: The Role of L-arginine in Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Prof., Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-arginine and PCOS
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrome; L-arginine; Gut Microbiome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- L-arginine intervention with 3g daily treatment for three months (Experimental): L-arginine therapy
  Interventions: Drug: L-arginine intervention

INTERVENTIONS:
Drug: L-arginine intervention — L-arginine intervention for 3 months, 3 g per day.

SUMMARY:
PCOS patients meeting the trial criteria were enrolled from the Shanghai 10th People's Hospital. The contents of this study were introduced to them, and they were invited to participate in the study. We further evaluated the efficacy and safety of arginine in treating PCOS by implementing the L-arginine clinical intervention protocol, and conducting post-intervention follow-up, efficacy evaluation, laboratory tests, and fecal sample 16S rRNA sequencing.

DETAILED DESCRIPTION:
In this study, we will enroll PCOS patients who meet the trial criteria from the Shanghai 10th People's Hospital, introduce the content of this study to them, and invite them to participate in the study. Perform laboratory tests for PCOS and collect baseline stool and blood samples. The clinical intervention program of L-arginine was implemented, and post-intervention follow-up, efficacy evaluation and laboratory examination were carried out. Stool and blood samples were collected after the intervention, and 16S rRNA sequencing was performed on stool samples before and after the intervention. To analyze whether PCOS-related clinical and laboratory indicators improved after L-arginine treatment of PCOS, and to analyze the changes in patients' microbiome before and after L-arginine treatment, to clarify the effectiveness and safety of L-arginine treatment of PCOS.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years
* Diagnosis of PCOS with the Rotterdam diagnosis criteria (2003)

Exclusion Criteria:

* Pregnant women;
* Hyperthyroidism or hypothyroidism
* Severe liver and kidney function injury
* Cancer patients;
* Associated with severe infection, severe anemia, neutropenia and other blood system diseases;
* Have type 1 diabetes, single-gene mutated diabetes or other secondary diabetes;
* Patients with mental illness or intellectual disability;
* Have a long history of taking hormone therapy;
* Currently or recently participating in another clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
menstrual frequency | Within 7 days of enrollment
  number of menstruation in a year

SECONDARY OUTCOMES:
Homeostasis model assessment of insulin resistance | Within 7 days of enrollment
  insulin resistance index
body mass index | Within 7 days of enrollment.
  body mass index (kg/m2)
fasting glucose | Within 7 days of enrollment.
  fasting glucose (mmol/L)
fasting insulin | Within 7 days of enrollment.
  fasting insulin (mmol/L)
Total cholesterol | Within 7 days of enrollment.
  Total cholesterol (mmol/L)
Triglycerides | Within 7 days of enrollment.
  Triglycerides (mmol/L)
HDL-c | Within 7 days of enrollment.
  HDL-c (mmol/L)
LDL-c | Within 7 days of enrollment.
  LDL-c (mmol/L)
total testosterone | Within 7 days of enrollment.
  total testosterone (nmol/L)
free testosterone | Within 7 days of enrollment.
  free testosterone (nmol/L)
Sex hormone-binding globulin | Within 7 days of enrollment.
  Sex hormone-binding globulin (nmol/L)
Androstenedione | Within 7 days of enrollment.
  Androstenedione (ng/ml)
Dehydroepiandrosterone | Within 7 days of enrollment.
  Dehydroepiandrosterone (ug/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Manna Zhang, doctor, Principal Investigator — Shanghai 10th People's Hospital
Locations (2):
- China (2):
  - Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No